CLINICAL TRIAL: NCT02811302
Title: PRediction of Opioid-induced Respiratory Depression In Patients Monitored by capnoGraphY (PRODIGY)
Brief Title: PRediction of Opioid-induced Respiratory Depression In Patients Monitored by capnoGraphY
Acronym: PRODIGY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: COVMOPO0560
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Results first posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-04

CONDITIONS: Respiratory Depression
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients monitored by capnography (Other): Capnography and pulse oximetry monitoring data will be collected for up to 48 hours while patients are on the hospital ward. In addition, a 1-month follow up will be completed.
  Interventions: Device: Capnostream Monitor

INTERVENTIONS:
Device: Capnostream Monitor — Capnography and pulse oximetry monitoring data will be collected for up to 48 hours while patients are on the hospital ward. In addition, a 1-month follow up will be completed.

SUMMARY:
PRODIGY is a prospective, multi-center, post-market, international cohort study. The primary objective of this study is to derive a score to identify subjects at risk to have respiratory depression (RD) episodes in patients undergoing opioid therapy in the hospital ward and monitored by capnography. The score will be derived by using subjects within the derivation cohort and internally validated using subjects within the validation cohort.

The primary endpoint used to derive the score will be the occurrence of RD episodes derived by Capnostream 20p device memory data combined with clinical data and validated by an independent Clinical Endpoint Committee (CEC) during the study course.

ELIGIBILITY:
Inclusion Criteria:

1. Patients receiving parenteral opioid therapy (for post-surgical or non-surgical) pain on the hospital ward.
2. Adult age (≥18 year old in US and Europe; ≥20 years old in Japan; ≥21 years old in Singapore).
3. Patient is able and willing to give informed consent.

Exclusion Criteria:

1. Expected length of stay ≤ 24 hours.
2. Patient is receiving intrathecal opioids.
3. Post-surgical patients with American Society of Anesthesiologists physical status (ASA PS) V or higher.
4. Patients with the status of Do Not Resuscitate (DNR), hospice, or receiving end of life therapy.
5. Ventilated or intubated patients.
6. Patient is unwilling or unable to comply fully with study procedures (including non-toleration of the capnography cannula) due to any disease condition which can raise doubt about compliance and influencing the study outcome.
7. Patient is a member of a vulnerable population, including legal incapacity or evidence that a subject cannot understand the purpose and risks of the study, regardless of authorized representative support.
8. Patient is participating in another potentially confounding drug or device clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1495 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2018-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank J Overdyk, Study Chair — Roper St. Francis Healthcare
Locations (16):
- United States (9):
  - University of Colorado Hospital, Aurora, Colorado
  - Emory University Hospital, Atlanta, Georgia
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - Buffalo General Medical Center, Buffalo, New York
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Providence Regional Medical Center Everett, Everett, Washington
- Hospital Foch, Suresnes, France
- University Hospital Bonn, Bonn, Germany
- Japan (2):
  - Okayama University Hospital, Okayama
  - The Jikei University School of Medicine Hospital, Tokyo
- Maastricht UMC+, Maastricht, Limburg, Netherlands
- National University Hospital, Singapore, Singapore
- Hospital Clínico Universitario de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Overdyk FJ, Carter R, Maddox RR, Callura J, Herrin AE, Henriquez C. Continuous oximetry/capnometry monitoring reveals frequent desaturation and bradypnea during patient-controlled analgesia. Anesth Analg. 2007 Aug;105(2):412-8. doi: 10.1213/01.ane.0000269489.26048.63. PMID 17646499
- [Background] Jarzyna D, Jungquist CR, Pasero C, Willens JS, Nisbet A, Oakes L, Dempsey SJ, Santangelo D, Polomano RC. American Society for Pain Management Nursing guidelines on monitoring for opioid-induced sedation and respiratory depression. Pain Manag Nurs. 2011 Sep;12(3):118-145.e10. doi: 10.1016/j.pmn.2011.06.008. PMID 21893302
- [Background] Cashman JN, Dolin SJ. Respiratory and haemodynamic effects of acute postoperative pain management: evidence from published data. Br J Anaesth. 2004 Aug;93(2):212-23. doi: 10.1093/bja/aeh180. Epub 2004 May 28. PMID 15169738
- [Background] Sun Z, Sessler DI, Dalton JE, Devereaux PJ, Shahinyan A, Naylor AJ, Hutcherson MT, Finnegan PS, Tandon V, Darvish-Kazem S, Chugh S, Alzayer H, Kurz A. Postoperative Hypoxemia Is Common and Persistent: A Prospective Blinded Observational Study. Anesth Analg. 2015 Sep;121(3):709-715. doi: 10.1213/ANE.0000000000000836. PMID 26287299
- [Derived] Doufas AG, Laporta ML, Driver CN, Di Piazza F, Scardapane M, Bergese SD, Urman RD, Khanna AK, Weingarten TN; Prediction of Opioid-induced respiratory Depression In patients monitored by capnoGraphY (PRODIGY) Group Investigators. Incidence of postoperative opioid-induced respiratory depression episodes in patients on room air or supplemental oxygen: a post-hoc analysis of the PRODIGY trial. BMC Anesthesiol. 2023 Oct 4;23(1):332. doi: 10.1186/s12871-023-02291-x. PMID 37794334
- [Derived] Kor JJ, Sprung J, Khanna AK, Weingarten TN. Continuous Monitoring Detected Respiratory Depressive Episodes in Proximity to Adverse Respiratory Events During the PRODIGY Trial. J Patient Saf. 2022 Dec 1;18(8):738-741. doi: 10.1097/PTS.0000000000001003. Epub 2022 Apr 27. PMID 35405725
- [Derived] Sim MA, Seet E, Khanna AK, Weingarten TN, Liew L, Law LS, Liu KE, Di Piazza F, Ti LK; PRediction of Opioid-induced respiratory Depression In patients monitored by capnoGraphY (PRODIGY) Group Investigators. Association Between Race and Opioid-Induced Respiratory Depression: An International Post Hoc Analysis of the Prediction of Opioid-induced Respiratory Depression In Patients Monitored by Capnography Trial. Anesth Analg. 2022 Nov 1;135(5):1097-1105. doi: 10.1213/ANE.0000000000006006. Epub 2022 Mar 29. PMID 35350054
- [Derived] Khanna AK, Jungquist CR, Buhre W, Soto R, Di Piazza F, Saager L; PRediction of Opioid-induced respiratory Depression In patients monitored by capnoGraphY (PRODIGY) Group Investigators. Modeling the Cost Savings of Continuous Pulse Oximetry and Capnography Monitoring of United States General Care Floor Patients Receiving Opioids Based on the PRODIGY Trial. Adv Ther. 2021 Jul;38(7):3745-3759. doi: 10.1007/s12325-021-01779-7. Epub 2021 May 24. PMID 34031858
- [Derived] Khanna AK, Saager L, Bergese SD, Jungquist CR, Morimatsu H, Uezono S, Ti LK, Soto R, Jiang W, Buhre W. Opioid-induced respiratory depression increases hospital costs and length of stay in patients recovering on the general care floor. BMC Anesthesiol. 2021 Mar 20;21(1):88. doi: 10.1186/s12871-021-01307-8. PMID 33743588
- [Derived] Urman RD, Khanna AK, Bergese SD, Buhre W, Wittmann M, Le Guen M, Overdyk FJ, Di Piazza F, Saager L. Postoperative opioid administration characteristics associated with opioid-induced respiratory depression: Results from the PRODIGY trial. J Clin Anesth. 2021 Jun;70:110167. doi: 10.1016/j.jclinane.2021.110167. Epub 2021 Jan 22. PMID 33493688
- [Derived] Khanna AK, Bergese SD, Jungquist CR, Morimatsu H, Uezono S, Lee S, Ti LK, Urman RD, McIntyre R Jr, Tornero C, Dahan A, Saager L, Weingarten TN, Wittmann M, Auckley D, Brazzi L, Le Guen M, Soto R, Schramm F, Ayad S, Kaw R, Di Stefano P, Sessler DI, Uribe A, Moll V, Dempsey SJ, Buhre W, Overdyk FJ; PRediction of Opioid-induced respiratory Depression In patients monitored by capnoGraphY (PRODIGY) Group Collaborators. Prediction of Opioid-Induced Respiratory Depression on Inpatient Wards Using Continuous Capnography and Oximetry: An International Prospective, Observational Trial. Anesth Analg. 2020 Oct;131(4):1012-1024. doi: 10.1213/ANE.0000000000004788. PMID 32925318
- [Derived] Khanna AK, Overdyk FJ, Greening C, Di Stefano P, Buhre WF. Respiratory depression in low acuity hospital settings-Seeking answers from the PRODIGY trial. J Crit Care. 2018 Oct;47:80-87. doi: 10.1016/j.jcrc.2018.06.014. Epub 2018 Jun 18. PMID 29936327

RESULTS

PARTICIPANT FLOW:
Groups:
- Full Analysis Set: Blinded capnography monitoring - all subjects enrolled
Period: Overall Study
Arm/Group | Full Analysis Set
Started | 1495
Completed | 1282
Not Completed | 213

BASELINE CHARACTERISTICS:
Population: Consented subjects that met eligibility criteria.
Groups:
- Single Cohort: Blinded capnography monitoring - all subjects enrolled
Arm/Group | Single Cohort
Number analyzed (Participants) | 1495
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 subject missing data
  Participants
    number analyzed (Participants) | 1494
    Female | 859
    Male | 635
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnic Origin: American Indian or Alaska Native | 5
  Race/Ethnic Origin: Asian | 325
  Race/Ethnic Origin: Black or African American | 174
  Race/Ethnic Origin: Hispanic or Latino | 10
  Race/Ethnic Origin: Native Hawaiian or Other Pacific Islander | 1
  Race/Ethnic Origin: Other | 36
  Race/Ethnic Origin: White | 839
  Race/Ethnic Origin: Missing Data | 105
Region of Enrollment [Number; unit: participants]
  Netherlands | 92
  Singapore | 100
  United States | 878
  Japan | 219
  France | 52
  Germany | 57
  Spain | 97
Weight [Mean (Standard Deviation); unit: kg] | 83.2 (25.2)
Height [Mean (Standard Deviation); unit: cm] | 167.1 (10.9)
Shirt Collar Neck Size [Count of Participants; unit: Participants]
  Male - shirt collar <17 in/43 cm | 377
  Male - shirt collar >= 17 in/43 cm | 221
  Female - shirt collar <16 in/41 cm | 561
  Female - shirt collar >=16 in/41 cm | 259
  Missing Data | 77
ASA Score [Count of Participants; unit: Participants] — Global anesthetic condition classification scale based upon health status assessment with range of ASA I (normal healthy patient) to ASA VI (declared brain dead patient whose organs are being removed for donor purposes). Multiple criteria are considering when assigning a physical status classification to a patient, such as smoking status, Body Mass Index, and medical history. Status was determined by the patient's surgical/anesthesia team. A higher score correlates to poorer outcomes.
  Participants
    Class I | 122
    Class II | 703
    Class III | 610
    Class IV | 33
    Missing Data | 27
Altitude [Count of Participants; unit: Participants]
  At or Below Sea Level | 72
  Above Sea Level to Below High Alititude | 1228
  High Altitude (1500-3500 meters) | 105
  Very High Altitude (above 3500 meters) | 3
  Missing Data | 87
STOP-BANG Score [Mean (Standard Deviation); unit: units on a scale] — The STOP-BANG score is a tool to determine if a patient is at risk for Obstructive Sleep Apnea (OSA). Parameters that are assessed include whether a person snores, is tired, has high blood pressure, or has been observed to stop breathing while asleep, has a Body Mass Index higher than 35 kg/m^2, age, gender, neck circumference. The score ranges from 0 to 8, and includes three risk categories for OSA (Low = 0-2, Intermediate = 3-4, High = 5-8).
  Chung F et al. Anesthesiology 2008; 108: 812-821, Chung F et al Br J Anaesth 2012; 108: 768-775, Chung F et al J Clin Sleep Med Sept 2014.
  units on a scale | 2.8 (1.7)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.7 (8.3)
Apnea History [Count of Participants; unit: Participants]
  Snore Loudly: Yes | 445
  Snore Loudly: No | 955
  Snore Loudly: Missing Data | 95
  Tired, Fatigued, Sleepy During the Day: Yes | 267
  Tired, Fatigued, Sleepy During the Day: No | 1132
  Tired, Fatigued, Sleepy During the Day: Missing Data | 96
  Stop Breathing or Choking/Gasping During Sleep: Yes | 152
  Stop Breathing or Choking/Gasping During Sleep: No | 1249
  Stop Breathing or Choking/Gasping During Sleep: Missing Data | 94
  Treated for High Blood Pressure: Yes | 678
  Treated for High Blood Pressure: No | 812
  Treated for High Blood Pressure: Missing Data | 5

OUTCOME MEASURES:

1. Primary Outcome: Determine Number of Subjects With RD While on Opioid Therapy
Description: Continuous respiratory monitoring using a Capnostream monitor will be included for collecting data for end tidal carbon dioxide (etCO2) and Oxygen saturation (SpO2). Positive RD determination was provided by an independent Clinical Event Committee, by assessing the following parameters:
  * etCO2 ≤ 15 or ≥ 60 mmHg for ≥ 3 minutes, or
  * RR ≤ 5 breaths for ≥ 3 minutes, or
  * SpO2 ≤ 85% for ≥ 3 minutes, or
  * Apnea episode lasting > 30 seconds, or
  * Any respiratory Opioid-Related Adverse Event (rORADE).
Time Frame: 48 hours
Population: A modified dataset (mFAS) was used to derive and validate the risk assessment tool. Subjects with major deviations or consent withdrawals; subjects which had no continuous monitoring data were also excluded. A total of 1336 patients were included in the derivation and validation of the tool.
Measure: Count of Participants; unit: Participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 1495
Participants
  RD | 655
  No RD | 840
Statistical Analysis 1: Comparison: Full Analysis Set; Test type: Other — A simple count and percentage of the population were calculated based on the number of patients adjudicated as having Respiratory Depression; To determine the risk assessment score, first the number of patients with Respiratory Depression (RD) had to be identified. Per the rules established for the Clinical Endpoint Committee, 655 (43.6%) patients were identified as having RD

2. Primary Outcome: To Derive and Validate a Risk Assessment Tool to Identify Subjects at Risk of Having RD While Undergoing Opioid Therapy on the Hospital Ward
Description: A risk assessment tool will be derived and validated using the incidence of RD episodes captured by continuous capnography and pulse oximetry measurements recorded on the Capnostream device memory data in conjunction with the clinical data as reported by the investigator.
Time Frame: 48 hours
Population: A modified dataset (mFAS) was used to derive and validate the risk assessment tool. Subjects excluded from the mFAS had major deviations or consent withdrawals or had no continuous monitoring data.
Measure: Count of Participants; unit: Participants
Groups:
- Full Analysis Dataset: All subjects enrolled
Arm/Group | Full Analysis Dataset
Number analyzed (Participants) | 1266
Participants
  Low Risk for RD | 351
  Intermediate Risk for RD | 457
  High Risk for RD | 458
Statistical Analysis 1: Comparison: Full Analysis Dataset; A modified Full Analysis Dataset (1335) was used to derive and validate the risk assessment tool. Subjects were excluded if they had major deviations or consent withdrawals. Subjects that did not have any monitoring data were also excluded. Finally, 69 subjects were further excluded from the model, as they were missing parameters to calculate their risk score; Test type: Other — Multivariable model for (Multivariate logistic regression) Respiratory Depression, followed by validation with Harrell's Optimism using a bootstrap sampling method; Area Under the Curve = 0.76, 95% CI 2-sided [0.73 to 0.79] — The model was performed using stepwise selection including all potential predictors and interactions terms (medical history and baseline characteristics); The model derived from the logistic regression was assessed by the Hosmer-Lemshow goodness of fit test (P = 0.831). The derived model was validated by Harrell's Optimism using a Bootstrap sampling method (500 samples from the modified dataset, 1335) with replacement. The logistic regression model with stepwise selection was performed for each bootstrap sample, and AUC calculated. The optimism calculated by Harrell's algorithm was 0.02. The model was then checked for the quartiles of the effective monitoring and for geography used as a random effect. The performance measurement of the final model was adjusted according the Harrell's Optimism for a final adjusted AUC of 0.74

ADVERSE EVENTS:
Time Frame: 1 month (+/- 10 days)
Description: ISO 14155:2001 definitions were applied to this study. Adverse Event rates for subjects with and without RD were characterized and compared. All subjects were considered in the Adverse Event evaluations (Full Analysis Dataset, 1495). Adverse Events were collecte if they had an underlying respiratory cause, was an adverse device effect (ADE) or was a Serious Adverse Event.
Groups:
- Blinded Capnography Monitoring: Subjects were clinically monitored through standard methods (standard clinical practice at the site), as well as with continuous data collection from the Capnostream monitor for a maximum of 48 hours. The monitoring period started for subjects once they arrived on the ward, for those subjects where opioid therapy was initiated prior to arrival on the hospital ward. Monitoring was permitted to be discontinued after a minimum of 4 hours from the last dose of opioid therapy received or if the subject was discharged from the hospital ward.
  No treatments were administered for this study. This study was observational in nature for all subjects. The capnography monitor served primarily as a data collection method. The capnography monitor screen was blinded, and alarms silenced for all subjects.
Arm/Group | Blinded Capnography Monitoring
All-Cause Mortality (participants affected / at risk) | 2/1495
Serious Adverse Events (participants affected / at risk) | 145/1495
Other Adverse Events (participants affected / at risk) | 181/1495
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blinded Capnography Monitoring (N=1495)
Arrythmia (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 2 (2)
Atrial Tachycardia (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
Pyloric Stenosis (Congenital, familial and genetic disorders) | 1 (1)
Abdominal Hernia (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 3 (3)
Ascites (Gastrointestinal disorders) | 1 (1)
Colitis Ulcerative (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Duodenal Ulcer (Gastrointestinal disorders) | 1 (1)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Wall Thickening (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 6 (6)
Impaired Gastric Emptying (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (1)
Peritoneal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 (2)
Subileus (Gastrointestinal disorders) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1) — Opioid related side effect
Chest Pain (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Systematic inflammatory response syndrome (General disorders) | 1 (1)
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 (1)
Portal Vein Thrombosis (Hepatobiliary disorders) | 1 (1)
Abdominal Abscess (Infections and infestations) | 1 (1)
Abdominal Infection (Infections and infestations) | 2 (2)
Abdominal wall abscess (Infections and infestations) | 1 (1)
Abscess (Infections and infestations) | 1 (1)
Abscess soft tissue (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Colonic Abscess (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 3 (3) — Hip Implants (2), PICC Line (1)
Incision Site Cellulitis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Perineal Abscess (Infections and infestations) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 8 (8)
Post Procedural Infection (Infections and infestations) | 1 (1)
Post Procedural Sepsis (Infections and infestations) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 6 (6)
Polynephritis Acute (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Sepsis Syndrome (Infections and infestations) | 1 (1)
Staphylococcal Infection (Infections and infestations) | 2 (2)
Stoma Site Cellulitis (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 2 (2)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1)
Wound Abscess (Infections and infestations) | 2 (2)
Wound Infection (Infections and infestations) | 2 (2)
Anastomotic complication (Injury, poisoning and procedural complications) | 1 (1)
Anastomotic lead (Injury, poisoning and procedural complications) | 2 (2)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Joint Dislocation (Injury, poisoning and procedural complications) | 3 (3)
Pancreatic Leak (Injury, poisoning and procedural complications) | 1 (1)
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 (1)
Post Procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 2 (2)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 2 (2)
Procedural Vomiting (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 2 (2)
Stoma Site ischaemia (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Wound Complication (Injury, poisoning and procedural complications) | 1 (1)
Wound evisceration (Injury, poisoning and procedural complications) | 1 (1)
Breath sounds abnormal (Investigations) | 1 (1)
Liver Function Test Abnormal (Investigations) | 1 (1)
Oxygen Saturation decreased (Investigations) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Investigations) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal instability (Musculoskeletal and connective tissue disorders) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Device Disclocation (Product Issues) | 2 (2) — Prostheses (2)
Delirium (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal Injury (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Colostomy closure (Surgical and medical procedures) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 1 (1)
Wound closure (Surgical and medical procedures) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blinded Capnography Monitoring (N=1495)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 17 (20)
Medical Device Discomfort (General disorders) | 167 (168)

LIMITATIONS AND CAVEATS:
Inconsistent reporting of opioid dosing frequency and amounts which led to the use of opioid naïve as a predictor, versus dose ranges. The scoring system should be further validated in a different study as an external validation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-11-29): https://cdn.clinicaltrials.gov/large-docs/02/NCT02811302/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/02/NCT02811302/SAP_001.pdf